CLINICAL TRIAL: NCT06968806
Title: Study on Ketorolac for Improving Outcomes and Prognosis in Patients With Stanford Type A Aortic Dissection -A Single-Center, Randomized, Double-Blind, Controlled Clinical Trial
Brief Title: Study on Ketorolac for Improving Outcomes and Prognosis in Patients With Stanford Type A Aortic Dissection
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); Huai'an First People's Hospital (Other); Shandong Provincial Hospital (Other Government); First Affiliated Hospital of Harbin Medical University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); THE FIRST AFFILIATED HOSPITAL OF SHIHEZI UNIVERSITY (Unknown); Xinhua Hospital of Ili Kazak Autonomous Prefecture (Unknown); Henan Provincial Chest Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025 -0039-02
Record Dates: First submitted 2025-03-31; First posted 2025-05-13 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-03

CONDITIONS: Aortic Dissection; Inflammation
Keywords: Inflammation; Aortic Dissection; Ketorolac
MeSH Terms: conditions — Aortic Dissection; Inflammation | interventions — Ketorolac; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: After enrollment, patients in the experimental group will receive ketorolac treatment for Stanford Type A aortic dissection, consisting of a 60mg intramuscular injection preoperatively followed by 30mg twice daily for two days postoperatively, while maintaining standard baseline therapies including analgesia, blood pressure control, and subsequent cardiovascular surgical management. The control group will receive identical placebo treatment (0.9% saline) with the same dosage regimen, formulation, and timing of administration as the experimental group, while also continuing all standard baseline treatments and surgical interventions without modification. Both groups will follow identical protocols except for the active drug versus placebo.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketorolac Group (Experimental): patients in the experimental group will receive ketorolac treatment for Stanford Type A aortic dissection, consisting of a 60mg intramuscular injection preoperatively followed by 30mg twice daily for two days postoperatively, while maintaining standard baseline therapies including analgesia, blood pressure control, and subsequent cardiovascular surgical management.
  Interventions: Drug: Ketorolac
- Placebo Group (Placebo Comparator): The control group will receive identical placebo treatment (normal saline) with the same dosage regimen, formulation, and timing of administration as the experimental group, while also continuing all standard baseline treatments and surgical interventions without modification. Both groups will follow identical protocols except for the active drug versus placebo
  Interventions: Drug: 0.9 % saline

INTERVENTIONS:
Drug: Ketorolac — patients in the experimental group will receive ketorolac treatment for Stanford Type A aortic dissection, consisting of a 60mg intramuscular injection preoperatively followed by 30mg twice daily for two days postoperatively, while maintaining standard baseline therapies including analgesia, blood pressure control, and subsequent cardiovascular surgical management.
  Arms: Ketorolac Group
Drug: 0.9 % saline — 0.9% saline
  Arms: Placebo Group

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled trial evaluates the efficacy and safety of ketorolac in 360 patients with Stanford Type A aortic dissection, conducted between 2025 and 2027. Participants will receive either ketorolac (60 mg intramuscularly [IM] preoperatively and 30 mg twice daily [BID] for two days postoperatively) or placebo in addition to standard care. Study outcomes include composite clinical endpoints, postoperative complications, and adverse events, which will be assessed through clinical evaluations, laboratory testing, and imaging studies at predefined intervals up to 90 days. The objective of this trial is to determine whether perioperative administration of ketorolac improves clinical outcomes in this patient population.

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind, controlled clinical trial will enroll 360 eligible patients with Stanford Type A aortic dissection between March 2025 and December 2027. Participants will be equally randomized to receive either ketorolac (intervention group: 60 mg intramuscular [IM] preoperatively followed by 30 mg twice daily [BID] for two days postoperatively) or matching placebo (control group), with both groups receiving standard perioperative care including analgesia, blood pressure control, and surgical treatment. Comprehensive data collection will include demographic characteristics, clinical parameters, laboratory tests (complete blood count [CBC], biochemistry, coagulation profile, cardiac enzymes, procalcitonin, cultures), and imaging studies (radiomics, biomechanics, chest X-ray, ultrasound, computed tomography [CT], magnetic resonance imaging [MRI]) at multiple timepoints from admission through 90-day follow-up. The primary outcomes will focus on evaluating the efficacy and safety of ketorolac through analysis of composite endpoint events, complication rates, and adverse reactions, with immediate study discontinuation and reporting for any treatment-related adverse events. All treatment protocols will maintain identical administration schedules and formulations between groups, with the exception of the active drug versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Stanford Type A aortic dissection confirmed by imaging and scheduled for emergency surgery.

Aged between 18 and 65 years.

Signed informed consent.

Exclusion Criteria:

* Patients who are unable to eat independently or require prolonged fasting.

History of malignant tumors.

Body weight <50 kg.

Traumatic aortic dissection.

Patients with Marfan syndrome.

Unstable vital signs requiring preoperative mechanical support or resuscitation (e.g., IABP [Intra-Aortic Balloon Pump], ECMO [Extracorporeal Membrane Oxygenation], LVAD [Left Ventricular Assist Device])

Patients requiring preoperative endotracheal intubation.

Consciousness impairment, central nervous system dysfunction, or evidence of cerebral malperfusion syndrome upon admission.

Preoperative hematemesis, melena, fresh blood in stool, or symptoms of bowel dilation.

Clear evidence of limb malperfusion before surgery.

Presence of organ malperfusion syndrome.

Patients requiring interventional procedures to relieve organ malperfusion before surgery.

History of gastrointestinal ulcers or chronic gastrointestinal inflammatory diseases.

History of dialysis or renal insufficiency before admission.

History of liver disease.

Allergy to ketorolac tromethamine, aspirin, or other nonsteroidal anti-inflammatory drugs (NSAIDs).

Chronic inflammatory diseases, autoimmune diseases, or long-term use of steroids or NSAIDs for other reasons.

Absence of cerebral perfusion during deep hypothermic circulatory arrest.

History of major surgery or acute myocardial infarction within 90 days.

History of cardiac or major vascular surgery.

Pregnant or lactating women.

Patients who refuse to participate in this clinical trial or decline to sign the informed consent form.

Any other conditions deemed unsuitable for participation by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Composite Endpoint: Mortality, Malperfusion Syndrome, Permanent Organ Dysfunction, Unplanned Cardiac Reoperation, and Prolonged Hospitalization | Continuous intervention for 3 days after admission, with a 1-year follow-up.
  The composite endpoint includes death (the worst outcome); malperfusion syndrome (including myocardial ischemia, stroke, lower limb paralysis, acute abdominal syndrome, renal failure requiring temporary dialysis, or symptoms and signs of limb ischemia); permanent dialysis, tracheostomy, or neurological deficits at discharge; postoperative mechanical circulatory support or unplanned cardiac reoperation (excluding reoperation for bleeding); postoperative cardiac arrest, multiple organ failure, or mechanical ventilation support for more than 72 hours; and postoperative hospital stay of 91 days or longer.

SECONDARY OUTCOMES:
erythrocyte sedimentation rate (ESR) | Preoperative and postoperative assessments on days 1, 3, 5, 7, 30, and 90
  erythrocyte sedimentation rate (ESR), an indicator of systemic inflammation that reflects the rate at which red blood cells settle in a vertical tube over a specified period. Elevated ESR levels may suggest ongoing inflammatory responses, infection, or tissue injury
The perioperative use of opioids | perioperative
  The perioperative use of opioids such as fentanyl and remifentanil is also assessed
C-reactive protein (CRP) | Preoperative and postoperative assessments on days 1, 3, 5, 7, 30, and 90
  C-reactive protein (CRP), an acute-phase protein synthesized by the liver that rises rapidly in response to infection, inflammation, or tissue injury. CRP serves as a sensitive biomarker of systemic inflammatory response and will be used to assess the perioperative inflammatory status in patients with Stanford Type A aortic dissection.
interleukin-6 (IL-6) | Preoperative and postoperative assessments on days 1, 3, 5, 7, 30, and 90
  interleukin-6 (IL-6), a pro-inflammatory cytokine produced by various cells in response to tissue injury, infection, or stress. IL-6 plays a key role in the acute-phase inflammatory response and is closely associated with the severity of systemic inflammation.
Complete Blood Count (CBC) | Preoperative and postoperative assessments on days 1, 3, 5, 7, 30, and 90
  A Complete Blood Count (CBC) is a common blood test that evaluates overall health and detects a wide range of disorders, including infections, anemia, and leukemia. It measures several components and features of the blood
Procalcitonin (PCT) | Preoperative and postoperative assessments on days 1, 3, 5, 7, 30, and 90
  Procalcitonin (PCT) is a protein precursor of the hormone calcitonin, which is involved in calcium metabolism. Normally, PCT is produced in the thyroid C cells and is present in very low levels in the blood. However, during severe bacterial infections, levels rise significantly, making it a useful biomarker for diagnosing and monitoring bacterial infections, sepsis, and guiding antibiotic therapy.
Prothrombin Time (PT) | Preoperative and postoperative assessments on days 1, 3, 5, 7, 30, and 90
  Prothrombin Time (PT) is a blood test that measures how long it takes for plasma to clot after adding thromboplastin (a reagent that activates the extrinsic pathway of coagulation). It evaluates the function of the extrinsic pathway (Factor VII) and common pathway (Factors X, V, II, and fibrinogen).
Activated Partial Thromboplastin Time (aPTT) | Preoperative and postoperative assessments on days 1, 3, 5, 7, 30, and 90
  Activated Partial Thromboplastin Time (aPTT) is a fundamental coagulation test that measures the time required for plasma to clot after activation of the intrinsic pathway. This test evaluates the functionality of all coagulation factors except Factor VII and XIII.
Platelet function | Preoperative and postoperative assessments on days 1, 3, 5, 7, 30, and 90
  Platelet function refers to the ability of platelets to participate in hemostasis through adhesion, activation, aggregation, and procoagulant activity. Proper platelet function is essential for primary hemostasis and vascular repair.
Alanine Aminotransferase (ALT) | Preoperative and postoperative assessments on days 1, 3, 5, 7, 30, and 90
  Alanine Aminotransferase (ALT), also known as serum glutamate-pyruvate transaminase (SGPT), is a liver enzyme primarily found in hepatocytes. It plays a key role in amino acid metabolism by catalyzing the transfer of an amino group from alanine to α-ketoglutarate, producing pyruvate and glutamate.
Creatinine | Preoperative and postoperative assessments on days 1, 3, 5, 7, 30, and 90
  Creatinine is a waste product generated from the breakdown of creatine phosphate in muscles. It is filtered by the kidneys and excreted in urine, making it a key marker for kidney function.
Creatine Kinase (CK) | Preoperative and postoperative assessments on days 1, 3, 5, 7, 30, and 90
  Creatine Kinase (CK), also known as Creatine Phosphokinase (CPK), is an enzyme that plays a critical role in cellular energy metabolism. It catalyzes the conversion of creatine + ATP ↔ phosphocreatine + ADP, providing rapid energy for muscle contraction.
Cardiopulmonary Bypass (CPB) Time | Intraoperative
  Cardiopulmonary Bypass (CPB) Time refers to the duration (in minutes) during which a patient's circulatory and respiratory functions are temporarily supported by a heart-lung machine during cardiac surgery. This allows surgeons to operate on a still, bloodless heart.
Total Surgical Duration | Intraoperative
  Total Surgical Duration refers to the entire time from skin incision to wound closure during a surgical procedure. It is a critical metric in perioperative medicine, influencing patient outcomes, resource utilization, and surgical team performance.
Postoperative drainage | Perioperative/Periprocedural
  Postoperative drainage refers to the fluid collected from surgical sites via drains, providing critical information about healing and complications. Monitoring its volume and characteristics helps guide clinical decisions.
Transfusion requirements | Perioperative/Periprocedural
  Transfusion requirements refer to the amount and type of blood products needed during or after surgery to maintain adequate oxygenation, hemostasis, and hemodynamic stability. The volume transfused depends on blood loss, preoperative anemia, and patient physiology.
Postoperative sternal infection (PSI) | Perioperative/Periprocedural
  Postoperative sternal infection (PSI) refers to surgical site infections involving the sternum after cardiac or thoracic surgery, particularly following median sternotomy. These infections range from superficial wound complications to life-threatening mediastinitis.
Number of Participants with breakthrough pain | Perioperative/Periprocedural
  Incidence: 20-40% of surgical patients experience inadequately controlled pain requiring rescue analgesia.
  Risk Factors:
  Major surgery (e.g., orthopedic, abdominal)
  Preoperative opioid use
  Younger age
Number of Participants with nausea | Perioperative/Periprocedural
  Nausea is an unpleasant, subjective sensation of impending vomiting, often accompanied by autonomic symptoms like pallor, sweating, and increased salivation. As a common postoperative complication, it represents a significant challenge in perioperative care.
Number of Participants with vomiting | Perioperative/Periprocedural
  Vomiting (emesis) is the forceful expulsion of gastric contents through the mouth resulting from coordinated contractions of the abdominal, thoracic, and gastrointestinal musculature. As a protective reflex mediated by the brainstem, it serves to eliminate harmful substances but becomes clinically significant when occurring postoperatively or pathologically.
Number of Participants with gastrointestinal discomfort | Perioperative/Periprocedural
  Gastrointestinal (GI) discomfort refers to a spectrum of subjective abdominal symptoms occurring postoperatively, distinct from nausea/vomiting. This nonspecific symptom complex affects 15-40% of surgical patients and significantly impacts recovery trajectories.
aortic tissue density | the 1-year follow-up
  imaging-based radiomics and biomechanical analyses from CTA and other modalities are used to evaluate aortic tissue density
aortic tissue strength | the 1-year follow-up
  maging-based radiomics and biomechanical analyses from CTA and other modalities are used to evaluate aortic tissue strength
abnormal blood flow | the 1-year follow-up
  imaging-based radiomics and biomechanical analyses from CTA and other modalities are used to evaluate abnormal blood flow
Survival rate | the 1-year follow-up
  Survival rate refers to the percentage of patients who remain alive for a specified period after diagnosis or treatment of a disease. It is a key metric in evaluating treatment efficacy, disease prognosis, and healthcare outcomes.
NYHA | he 1-year follow-up
  NYHA classification is a widely used system to categorize the severity of heart failure symptoms based on a patient's physical limitations. It helps clinicians assess disease progression, guide treatment decisions, and predict outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Tuo Pan, MD, Study Director — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; DongJin Wang, MD, Study Chair — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; DongJin Wang, MD, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No